CLINICAL TRIAL: NCT03334188
Title: A Clinical Trial of an Electronic Health Record-leveraged, Patient-centered, Intensification of Chronic Care for Heart Failure (EPIC-HF)
Brief Title: Electronic Health Record-leveraged, Patient-centered, Intensification of Chronic Care for HF
Acronym: EPIC-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-1249
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Results first posted 2021-09-17 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Patient Engagement; Medication Optimization; Heart Failure With Reduced Ejection Fraction; Patient Activation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Patients will receive care-as-usual. The only study procedures patients will be exposed to will be a baseline survey at time of enrollment about their sense of engagement around their HFrEF medication prescribing, as well as a follow-up survey with the same general content one month after their next clinic appointment. Medical record review will occur at baseline (enrollment), 1 month after the next clinic appointment post-enrollment, and at 12 months from enrollment.This arm will include 'No Intervention--Usual Care'.
  Interventions: Behavioral: No Intervention--Usual Care
- Intervention (Active Comparator): Patients will receive the patient engagement video and HFrEF medication checklist by email one week prior to their next clinic appointment after enrollment. Patients in the intervention arm will also receive a baseline survey at time of enrollment about their sense of engagement around their HFrEF medication prescribing, as well as a follow-up survey with the same general content one month after their next clinic appointment. Medical record review will occur at baseline (enrollment), 1 month after the next clinic appointment post-enrollment, and at 12 months from enrollment. This arm will include the 'Intervention :Behavioral: Patient engagement materials.'
  Interventions: Behavioral: Patient engagement materials

INTERVENTIONS:
Behavioral: Patient engagement materials — The intervention is a brief, animated video designed to engage and activate patients around their HFrEF medication prescribing, as well as a HFrEF medication checklist.
  Arms: Intervention
Behavioral: No Intervention--Usual Care — Control for intervention--patient receives care as usual from provider to contrast against intervention arm.
  Arms: Control

SUMMARY:
The EPIC-HF study will test the effectiveness of a patient empowerment and activation for optimization of Heart Failure with reduced Ejection Fraction (HFrEF) medication plans. Three main regional centers in the University of Colorado Health (UCHealth) system will participate in a two-arm, randomized study design. In this design, each site participates in both control and intervention, with members of the sites eligible patient population randomly enrolled in either the intervention or the control arm. All eligible patients who agree to participate in the study will complete the Baseline Survey, the Follow-Up Survey, and will have information collected from their medical record at baseline, 1 month after the first clinic appointment post-enrollment, and 1 year after enrollment. Enrollment will take place at three UCHealth locations: UCHealth University of Colorado Hospital (Metro), UCHealth Medical Center of the Rockies and UCHealth Poudre Valley Hospital (North), and UCHealth Memorial Central and Memorial North (South). Study personnel at the North and South sites will carry out enrollment and Baseline Surveys with patients for those locations; all other study procedures will be conducted by study personnel at the University of Colorado (UC) School of Medicine (SOM) (UCSOM) at UCHealth University of Colorado School of Medicine.

Patients enrolled in the intervention arm will receive, by email and/or text, a link to 1) a short patient engagement video around HFrEF medications, and 2) a link to an online portable document format (PDF) of a HFrEF medication checklist. Patients in the intervention arm will receive these materials after enrollment and one week prior to their next scheduled clinic appointment. The materials will be delivered in a second communication, three days after the first, via text, as well as a third communication on the day of the clinic appointment. Patients enrolled in the control arm will not receive any materials at any point of time and will receive their usual care.

For both arms, medication changes in patient medical records will be assessed before and after clinic visits to measure the effectiveness of the intervention on aim 1; surveys will be compared before and after clinic visits to determine the effectiveness of the intervention on aim 2.

DETAILED DESCRIPTION:
Multiple medications improve left ventricular remodeling, quality of life, and survival in patients with heart failure with reduced ejection fraction (HFrEF). Unfortunately, the real-world use of HFrEF medications is suboptimal, particularly for more recently approved agents such as aldosterone antagonists. The introduction of sacubitril/valsartan and ivabradine add to already complex HFrEF treatment regimens. Without novel mechanisms to improve medication use, the benefits of advances in HF treatment will be largely unrealized.

Efforts to optimize HFrEF medication delivery have focused primarily on 1) provider decision support around prescribing and 2) patient education around adherence. An important gap is the failure to empower patients to engage more directly in HFrEF prescribing efforts. Patients have a direct stake in making sure they are getting efficacious treatments, want to be involved in decisions about their treatments, and if engaged are more likely to adhere to them. Direct-to-consumer marketing and proliferation of shared decision making reflect a culture where patients are increasingly involved in medication prescribing.

Within this context, the American Heart Association (AHA) has funded four centers across the United States to examine ways in which heart failure treatment and prevention may be optimized. The University of Colorado, Denver is one of these sites; The Development and Trial of an Electronic health record-leveraged, Patient-centered, Intensification of Chronic care for Heart Failure Tool (EPIC-HF) is the population-focused arm of study. Inspired by the gap in HFrEF medication optimization, this study aims to develop a patient-centered intervention in order to 1) activate and engage patients with HFrEF in their prescribing regimen, 2) empower them to initiate discussions with their provider about ways in which their medication plan could be improved, which will result in 3) a superior HFrEF medication plan. The investigators modeled this tool with the previous success of flipped classrooms and patient empowerment initiatives in mind. The intervention was iteratively developed with the input of both clinician and patient stakeholders, and is innovative in its emphasis on patient self-actualization and role as an equal with their healthcare provider in the discussion around medication prescribing. This study applies the intervention in a two-arm, randomized controlled trial across three sites (UCHealth metro, Memorial, and Medical Center of the Rockies) in the UCHealth medical system.

Aim 1: Assess the effectiveness of the EPIC-HF intervention on HFrEF medication optimization Hypothesis 1: Compared to usual care, EPIC-HF will increase the number of HFrEF medication optimizations (i.e., dose changes for beta-blockers (βB), Angiotensin-converting enzyme inhibitors (ACE-I)/Angiotensin receptor blockers (ARB)/sacubitril, Aldosterone Receptor Antagonists (AldaA), Ivabradine, etc.) without compromising secondary outcomes including safety and healthcare provider satisfaction.

Aim 2: Assess the effectiveness of the EPIC-HF intervention on patient empowerment and activation around their HFrEF medication plan Hypothesis 2: Compared to usual care, EPIC-HF will result in increased patient empowerment and activation around their HFrEF medication plan as measured through patient self-assessment

ELIGIBILITY:
Inclusion Criteria:

1. Most recent cardiology imaging study showing left ventricular ejection fraction (LVEF) <=40%
2. A plan for ambulatory clinic appointments in the UCHealth system

Exclusion Criteria:

1. Patients who have clinic appointments more than 12 months apart
2. Under 18 years of age
3. Non-English speaking (decision tools and study assessments are in English only)
4. Unable to consent (this would include patients with conditions such as moderate-to- severe dementia)
5. Prisoners
6. Patients who are enrolled in hospice (increasing curative medications is often not appropriate in these patients)
7. Patients who are expected to live < 6 months as documented in the patient's chart by treating clinician.
8. Continuous IV inotropic support (e.g. dobutamine or milrinone)
9. Glomerular filtration rate (GFR) < 15 mL/min or chronic renal disease
10. Patients who have neither an email address nor a phone to which text messages may be sent
11. Patients with an left ventricular assist device (LVAD) implant
12. Patients who have neither an email address nor a phone to which text messages may be sent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Allen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allen LA, Venechuk G, McIlvennan CK, Page RL 2nd, Knoepke CE, Helmkamp LJ, Khazanie P, Peterson PN, Pierce K, Harger G, Thompson JS, Dow TJ, Richards L, Huang J, Strader JR, Trinkley KE, Kao DP, Magid DJ, Buttrick PM, Matlock DD. An Electronically Delivered Patient-Activation Tool for Intensification of Medications for Chronic Heart Failure With Reduced Ejection Fraction: The EPIC-HF Trial. Circulation. 2021 Feb 2;143(5):427-437. doi: 10.1161/CIRCULATIONAHA.120.051863. Epub 2020 Nov 17. PMID 33201741
- [Derived] Venechuk GE, Khazanie P, Page RL 2nd, Knoepke CE, Helmkamp LJ, Peterson PN, Pierce K, Thompson JS, Huang J, Strader JR, Dow TJ, Richards L, Trinkley KE, Kao DP, McIlvennan CK, Magid DJ, Buttrick PM, Matlock DD, Allen LA. An Electronically delivered, Patient-activation tool for Intensification of medications for Chronic Heart Failure with reduced ejection fraction: Rationale and design of the EPIC-HF trial. Am Heart J. 2020 Nov;229:144-155. doi: 10.1016/j.ahj.2020.08.013. Epub 2020 Aug 28. PMID 32866454

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Patients will receive care-as-usual. The only study procedures patients will be exposed to will be a baseline survey at time of enrollment about their sense of engagement around their heart failure with a reduced ejection fraction (HFrEF) medication prescribing, as well as a follow-up survey with the same general content one month after their next clinic appointment. Medical record review will occur at baseline (enrollment), 1 month after the next clinic appointment post-enrollment, and at 12 months from enrollment. This arm will include 'No Intervention--Usual Care'.
  No Intervention--Usual Care: Control for intervention--patient receives care as usual from provider to contrast against intervention arm.
- Intervention: Patients will receive the patient engagement video and HFrEF medication checklist by email one week prior to their next clinic appointment after enrollment. Patients in the intervention arm will also receive a baseline survey at time of enrollment about their sense of engagement around their heart failure with a reduced ejection fraction (HFrEF) medication prescribing, as well as a follow-up survey with the same general content one month after their next clinic appointment. Medical record review will occur at baseline (enrollment), 1 month after the next clinic appointment post-enrollment, and at 12 months from enrollment. This arm will include the 'Intervention :Behavioral: Patient engagement materials.'
  Patient engagement materials: The intervention is a brief, animated video designed to engage and activate patients around their HFrEF medication prescribing, as well as a HFrEF medication checklist.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 153 | 153
Completed | 145 | 145
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 1 | 0
Not completed — Never had qualifying clinic visit | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 145 | 145 | 290
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 64 [55 to 72] | 66 [58 to 74] | 65 [56.5 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 102 | 104 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 136 | 134 | 270
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 120 | 119 | 239
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 4 | 5 | 9
Employment [Count of Participants; unit: Participants]
  Employed | 45 | 46 | 91
  Retired | 59 | 72 | 131
  Unemployed | 39 | 23 | 62
  Missing | 2 | 4 | 6
Insurance [Count of Participants; unit: Participants]
  Medicare, Tricare | 71 | 73 | 144
  Medicaid | 23 | 21 | 44
  Private | 48 | 48 | 96
  None | 3 | 3 | 6
Income [Count of Participants; unit: Participants]
  Less than or equal to $20,000 | 31 | 24 | 55
  $20,001--$40,000 | 31 | 17 | 48
  $40,001--$60,000 | 15 | 20 | 35
  $60,001--$80,000 | 27 | 29 | 56
  Greater than $80,000 | 32 | 44 | 76
  Missing | 9 | 11 | 20
Single Relationship Status [Count of Participants; unit: Participants] | 59 | 56 | 115
Can receive text messages [Count of Participants; unit: Participants] | 86 | 77 | 163
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 110 [102 to 124] | 112.5 [104 to 124] | 111.3 [103 to 124]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 70 [62 to 80] | 70 [64 to 78] | 70 [63 to 79]
Pulse [Median (Inter-Quartile Range); unit: bpm (beats per minute)] | 74.5 [65.5 to 83] | 72.5 [68 to 80] | 73.5 [66.8 to 81.5]
left ventricular ejection fraction (LVEF) [Median (Inter-Quartile Range); unit: percent] | 32.5 [27 to 37.5] | 32.5 [25.2 to 37.5] | 32.5 [26 to 37.5]
brain natriuretic peptide (BNP) [Median (Inter-Quartile Range); unit: pg/mL] | 266 [126 to 728] | 161.5 [90 to 444.5] | 213.8 [108 to 586.3]
Serum creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.1 [0.9 to 1.4] | 1.0 [0.9 to 1.2] | 1.05 [0.9 to 1.3]
Serum potassium [Median (Inter-Quartile Range); unit: mmol/L] | 4.3 [3.9 to 4.6] | 4.2 [4.0 to 4.5] | 4.25 [3.95 to 4.55]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Experienced an Initiation or Intensification of Their Guideline-Directed Medical Therapy (GDMT)
Description: The investigators were interested in whether the patient engagement tool led to an increase in the optimization of HFrEF medications for patients. This was measured through medical record review of all medications and doses immediately preceding the cardiology clinic visit (enrollment) to 30 days after enrollment.
Time Frame: Enrollment, 1 month (30 days) after enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 145 | 145
percentage of participants | 29.7 | 49.0

2. Secondary Outcome: Self-Reported Patient Engagement Around HFrEF Medications
Description: The investigators were interested in whether the patient engagement tool (a 3-minute video and 1-page checklist-delivered electronically 1 week prior, 3 days prior and 24 hours prior to the enrollment cardiology clinic visit) led to an increase in patient sense of engagement around their HFrEF medication prescribing, prompting patients to begin a dialogue with their clinician about their medication plan. This was assessed among the Intervention group by comparing answers from a self-reported survey at 1 month after delivery of intervention materials. Participants were sent the survey and asked if they received and reviewed the intervention materials. Survey measures were included as well as a series of questions asking about how and when medications were discussed during clinical interactions.
Time Frame: 1 month after delivery of intervention materials.
Population: Of the 145 intervention patients that were sent the survey, 126 responded to the survey. Only intervention participants were analyzed for this outcome, since Control participants received usual care.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention - Only: Patients will receive the patient engagement video and HFrEF medication checklist by email one week prior to their next clinic appointment after enrollment. Patients in the intervention arm will also receive a baseline survey at time of enrollment about their sense of engagement around their HFrEF medication prescribing, as well as a follow-up survey with the same general content one month after their next clinic appointment. Medical record review will occur at baseline (enrollment), 1 month after the next clinic appointment post-enrollment, and at 12 months from enrollment. This arm will include the 'Intervention :Behavioral: Patient engagement materials.'
  Patient engagement materials: The intervention is a brief, animated video designed to engage and activate patients around their HFrEF medication prescribing, as well as a HFrEF medication checklist.
Arm/Group | Intervention - Only
Number analyzed (Participants) | 126
Participants
  Reported receiving the video | 81
  Reported reviewing the video | 73
  Found the video helpful in understanding their medical plan | 53
  Found the video helpful in discussing their medicines with their doctor | 51
  Reported receiving the checklist | 83
  Reported reviewing the checklist | 74
  Found the checklist helpful in understanding their medical plan | 56
  Found the checklist helpful in discussing their medicines with their doctor | 48
  Brought the checklist to their appointment | 61
  Talked about checklist with doctor at their appointment | 52

3. Secondary Outcome: Number of Participants With Initiation/Intensification of Key Heart Failure Medications
Description: Initiation or intensification of key heart failure medications was determined by medical chart review conducted at immediately following the cardiology clinic appointment (enrollment) and for the clinic visit closest to 1 month (30 days) after the enrollment visit. Raw numbers of participants were analyzed.
Time Frame: Enrollment, 1 month (30 days) after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 145 | 145
Participants
  Intensification occurring during cardiology clinic visit (day 1) | 42 | 61
  Any intensification in HFrEF medication, including GDMT, loop diuretic, or digoxin | 45 | 73
  Key heart failure medication added | 10 | 17
  Beta blocker added | 2 | 0
  ACE-I added | 1 | 4
  ARB added | 4 | 2
  ARNI added | 0 | 0
  Loop diuretic added | 0 | 0
  Aldosterone antagonist added | 3 | 5
  Ivabradine added | 0 | 1
  Hydralazine added | 1 | 1
  Isosorbide added | 1 | 2
  Digoxin added | 0 | 0
  ACE-I or ARB replaced with ARNI | 3 | 4
  Key heart failure medication up titrated | 33 | 58
  Beta blocker up titrated | 16 | 32
  ACE-I up titrated | 4 | 7
  ARB up titrated | 7 | 7
  ARNI up titrated | 5 | 6
  Loop diuretic up titrated | 1 | 0
  Aldosterone antagonist up titrated | 3 | 8
  Ivabradine up titrated | 0 | 0
  Hydralazine up titrated | 0 | 2
  Isosorbide up titrated | 0 | 1
  Digoxin up titrated | 0 | 0

4. Secondary Outcome: Guideline-directed Medical Therapy (GDMT) Intensifications Per Patient
Description: Guideline-directed medical therapy (GDMT) intensifications per patient from the pre-clinic visit (enrollment) to 1-month (30 days) after enrollment. This was measured by medical chart reviewing of the pre-clinic visit appointment and the closest clinic appointment preceding the 30 day mark after enrollment.
  Key: guideline directed medical therapy (GDMT); evidence-based beta blocker (EVBB); angiotensin converting enzyme inhibitors (ACE-I); angiotensin receptor blockers (ARB); angiotensin receptor neprilysin inhibitors (ARNI); mineralocorticoid receptor agonists (MRA); hydralazine/isosorbide dinitrate (H/ISDN); Ivabradine (Iva)
Time Frame: Enrollment, 1 month (30 days) after enrollment
Measure: Mean (Standard Deviation); unit: intensifications
Arm/Group | Control | Intervention
Number analyzed (Participants) | 145 | 145
intensifications
  # of GDMT intensifications (initiation/dose increase EVBB, ACEI, ARB, ARNI, MRA, H/ISDN, or Iva) | 0.36 (0.61) | 0.61 (0.73)
  # of all intensifications (including GDMT plus initiation or uptitration of loop diuretic or digoxin | 0.38 (0.62) | 0.63 (0.73)

5. Secondary Outcome: Safety Outcomes
Description: Unplanned hospitalizations or emergency department visits without hospitalization from the cardiology clinic visit (enrollment) to 1-month (30 days) after enrollment. Hospitalization and emergency department visits were obtained via medical chart review and were analyzed as yes/no per patient.
Time Frame: Enrollment, 1-month (30 days) after Enrollment
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 145 | 145
participants
  Unplanned hospitalization at 30 days | 4 | 6
  Emergency department visit without hospitalization at 30 days | 5 | 9

ADVERSE EVENTS:
Time Frame: 1 month (30 days) from Enrollment
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 1/145 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/145
Other Adverse Events (participants affected / at risk) | 0/145 | 0/145

LIMITATIONS AND CAVEATS:
We did not measure intolerance and contraindications to GDMT. Randomization occurred at the patient-level rather than the clinician- or site-level, which allowed for potential contamination. Only cardiology specialists were included in this study. The use of a single, regional health system may further limit generalizability. However University of Colorado Health is a diverse system spanning a range of local care approaches, and we over-enrolled under-represented patient groups where possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT03334188/Prot_SAP_000.pdf